CLINICAL TRIAL: NCT00739518
Title: Refinement and Assessment of New Magnetic Resonance Imaging (MRI) Technologies
Brief Title: Refinement and Assessment of New Magnetic Resonance Imaging Technologies for Neurological Exams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: General Electric (Industry); Philips Medical Systems (Industry)
Responsible Party: Principal Investigator, Ashok Srinivasan, M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00041731
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Nervous System Diseases
Keywords: Neurological; MRI
MeSH Terms: conditions — Nervous System Diseases; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI scan - new technology (Experimental): The patient's clinical MRI scan will also utilize some new technology, such as a change in software or additional MRI sequences
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Neurological MRI with new technology evaluation. The new technology may involve software or MRI scanning sequences. This is a long term research study that focuses on new technology that is constantly being created.

SUMMARY:
This study is being done to assess new Magnetic Resonance Imaging (MRI) technologies such as new hardware or software designed to improve MRI examinations of the brain, spine head and neck regions.

DETAILED DESCRIPTION:
This study is being done to assess new Magnetic Resonance Imaging (MRI) technologies such as new hardware or software designed to improve MRI examinations of the brain, spine, and head & neck regions.

Software and hardware are constantly being improved, new machines replace old machines, software is updated and improved as are the devices used to produce better MRI images.

ELIGIBILITY:
Inclusion Criteria:

* If you are a male or a non-pregnant female patient
* Normal volunteer
* presenting to MRI for a clinically-ordered neurological or head and neck MRI exam

Exclusion Criteria:

* Patients, who have electrically, magnetically or mechanically activated implants such as heart pacemaker, magnetic surgical clips, prostheses or implanted neurological stimulator.
* Pregnant patients or patients who are lactating.
* A patient who is claustrophobic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2004-10 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Improvement in quality of MRI studies in Neuroradiology | 1 year
  Specific Measurement Are:
  1. Scan speed - is the new method as fast or faster than regular method(s)
  2. Signal to noise - Subjectively, or quantitatively do we get the same, better, or new contrast compared to the regular methods(s).
  3. Image contrast - Subjectively, or quantitatively do we get the same or better resolution compared to the regular method(s).
  4. Spatial resolution - Subjectively, or quantitatively do we get the same or better resolution compared to the regular method(s).
  5. Artifact - Subjectively, or quantitatively do we get the better artifact reduction compared to the regular method(s).
  6. Ergonomics - Is the new software easier to work or offer more information more cleanly than the regular software
  7. Patient comfort - Subjectively, does the new software and/or hardware make the patient's MRI experience more comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Srivinasan, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No